CLINICAL TRIAL: NCT01534741
Title: Investigation on the Middle Size Molecule Elimination Characteristics of the FX CorDiax 60 in Relation to the FX 60-Dialyzer
Brief Title: Comparison FX CorDiax 60 in Relation to the FX 60-Dialyzer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Francisco Maduell, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HD-IIT-02-E
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2012-07

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Kidneys, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialyser (Active Comparator): FX CorDiax 60 dialyzer
  Interventions: Other: dialyzer comparison; Device: Dialyzer
- FXDialyser (Active Comparator): FX 60 dialyzer
  Interventions: Device: Dialyzer

INTERVENTIONS:
Other: dialyzer comparison — Each patient will be treated by post-dilution online hemodiafiltration once with each dialyzer type (FX CorDiax 60or FX 60 ) The order of dialyzers used will be randomly assigned to the patient at the time of randomisation by lot. Every subject will be treated one time with each dialyzer. In order to achieve controlled conditions, the mid- or end-week session data will be used, only.
  Arms: Dialyser
Device: Dialyzer — Comparison Dialyzer FX60 versus Cordiax60

SUMMARY:
Study design: Open, randomized, cross-over, monocentric, controlled, prospective Applied Medical Devices: FX CorDiax 60 (high-flux), FX 60 (high-flux) Patients: 30 adult chronic hemodialysis patients Treatment: Each patient will be treated by post-dilution online hemodiafiltration once with each dialyzer type.

Study objectives: Intraindividual comparison of removal rate of urea, phosphate, ß2-microglobulin (ß2-m), myoglobin, prolactin, alpha1-microglobulin and alpha1-acidglycoprotein and of the albumin loss with different dialyzer membranes during post-dilution online hemodiafiltration.

Primary variable: Removal rate of myoglobin Secondary variable: Removal rate of urea, phosphate, ß2-microglobulin (ß2-m), prolactin, alpha1-microglobulin and alpha1-acidglycoprotein Safety variable: Hematocrit, albumin loss Sample Size: 30 subjects

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated by post dilution on-line HDF for at least three months.
* Patients who reached a dialysis dose (Kt/V) of at least 1.2 at the last two monthly checks,
* Patients who are on a stable anticoagulation and anemia management,
* Patients who are clinically stable outlined by the medical history of the patient, based on judgment of principal investigator,
* Patients who are on a regular thrice weekly HDF schedule,
* Patients who have a good vascular access (fistula or graft) which enables easy insertion of the needles and suitable effective blood flow (> 300 ml/min),
* Patients who are able to understand the nature and requirements of the clinical investigation and have given written informed consent,
* Patients who are aged 18 years or older.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria,
* Patients with active HBV, HCV, HIV infection,
* Patients who are severely malnourished patients as judged by the principal investigator,
* Patients who are known or suspected to have allergy to the trial products or related products,
* Patients who are abusing non-legal drugs or alcohol (defined as an average daily intake of more than one liter of beer per day or an equivalent amount of alcohol in other beverages),
* Patients who have been diagnosed a current active malignant disease,
* Patients who participate simultaneously in another clinical investigation or in other clinical investigations during the last month,
* Patients who are uncooperative.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Removal rate of myoglobin | 2 weeks

SECONDARY OUTCOMES:
Removal rate of urea | 2 weeks
Removal rate of phosphate | 2 weeks
Removal rate of ß2-microglobulin (ß2-m) | 2 weeks
Removal rate of prolactin | 2 weeeks
Removal rate of alpha1-microglobulin | 2 weeks
Removal rate of alpha1-acid glycoprotein | 2 weeks
Hematocrit pre and post-dialysis | 2 weeks
Albumin loss during dialysis session | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Maduell F, Arias-Guillen M, Fontsere N, Ojeda R, Rico N, Vera M, Elena M, Bedini JL, Wieneke P, Campistol JM. Elimination of large uremic toxins by a dialyzer specifically designed for high-volume convective therapies. Blood Purif. 2014;37(2):125-30. doi: 10.1159/000358214. Epub 2014 Mar 20. PMID 24662288